CLINICAL TRIAL: NCT07370792
Title: CARTOGEN-N_Contribution of Optical Genome Mapping (OGM) in the Diagnosis of Multiple Congenital Malformations With or Without Intellectual Disability Without Genetic Abnormality Detected by Whole Genome Sequencing
Brief Title: Contribution of Optical Genome Mapping (OGM) in the Diagnosis of Multiple Congenital Malformations With or Without Intellectual Disability Without Genetic Abnormality
Acronym: CARTOGEN-N
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Céline PEBREL-RICHARD (Other)
Responsible Party: Sponsor-Investigator, Céline PEBREL-RICHARD, Dr, University Hospital, Clermont-Ferrand
Organization: University Hospital, Clermont-Ferrand (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOI 2024 PEBREL-RICHARD
Record Dates: First submitted 2025-12-09; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Congenital Malformations
Keywords: multiple congenital anomalies; non-contributive whole-genome sequencing; optical genome mapping; structural variants; genetic diagnosis
MeSH Terms: conditions — Congenital Abnormalities; Abnormalities, Multiple | interventions — Blood Specimen Collection

STUDY DESIGN:
Masking Description: Each sample will be pseudonymized as follows:
  CARTOGEN_N[patient number]-[initial of last name]-[initial of first name] Example: Pierre MARTIN, 15th enrolled patient → CARTOGEN_N[15]-[M]-[P]
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm of patients with congenital malformations (Experimental)
  Interventions: Genetic: blood sample

INTERVENTIONS:
Genetic: blood sample — A blood sample will be collected after obtaining consent from the patient and/or their legal guardians. The number of tubes required (1 to 3) will be determined according to the patient's weight, for the purpose of performing optical genome mapping and any necessary confirmatory analyses in the event that a structural variant is identified.

SUMMARY:
Congenital malformations result from an embryonic or foetal developmental disorder (DD) affecting one or more systems (cardiac, skeletal, nervous, etc.). These are referred to as multiple congenital anomalies (MCAs). They may be associated with an intellectual disability (ID)1.

Chromosomal analysis on Chromosomal Microarray Analysis (CMA) and gene panels or exome sequencing are the respective gold standard methods for chromosomal and molecular diagnosis of DD respectively2. In cases where no diagnosis is established after these first-line tests, short-read whole genome sequencing (WGS), via the Plan France Medicine Genomic 2020-2025 (AURAGEN), may be considered. This approach allows for diagnosis in nearly 40% of patients with DD3,4. However, many patients remain in diagnostic deadlock, likely due to the technical limitations of these methods, which potentially be overcome by emerging methodologies such as optical genome mapping (OGM)5,6,7,8,9. The investigators propose to systematically perform OGM in 30 patients presenting with MCA+/-ID who have inconclusive WGS result10.

The main objective is to assess the contribution of OGM in identifying structural variants not detected or poorly characterised by WGS in this clinical context. This work will also contribute to the ongoing of OGM in routine diagnostics and determine its role in the overall genetic diagnosis of MCA+/-ID. Additionally it may lead to the identification of new candidate genes and/or mechanisms of pathogenicity. If the results are promising, further clinical could expand this preliminary work into a larger-scale project. Improving the genetic diagnosis of DD should enhance the medical management of patients, currently in diagnostic deadlock, and their families.

DETAILED DESCRIPTION:
Study Workflow

Pre-analytical Phase

Participation in the study will be offered to all patients meeting the inclusion and non-inclusion criteria by an investigator from the Department of Genetics, during a medical consultation in which the non-contributive whole-genome sequencing (WGS) result will have been communicated (Figure 1). Information regarding the study procedures and objectives will be provided at that time. The information sheet and consent form will be given to the patient (if an adult) or to the holders of parental authority (if the patient is a minor). After obtaining consent for both the genetic investigations and participation in the research project, the patient may be enrolled in the study. Blood samples required for the study will be collected, transferred to the laboratory, and secured for analysis according to the following protocol:

Patient > 20 kg:

2 × 5 mL EDTA blood tubes

1. × 5 mL heparinized blood tube

   Patient 12-20 kg:
2. × 5 mL EDTA blood tubes

Patient 5-12 kg:

1 × 5 mL EDTA blood tube

Samples will be sent to the Cytogenetics Department, where they will be pseudonymized and secured. At least three aliquots of 1.5 mL EDTA blood and the remaining volume will be frozen at -80 °C for DNA extraction and long-fragment DNA extraction. A cell culture (peripheral blood lymphocytes) will also be performed to obtain a fixed chromosomal pellet from the heparinized tube, when available. If the heparinized sample is not available and the results of optical genome mapping require confirmation of a chromosomal abnormality by karyotype or FISH (i.e., contributive result), a second blood draw will be proposed during the clinical results-return consultation.

Analysis Frozen samples from the Cytogenetics Department of Clermont-Ferrand University Hospital (one per patient) will be transferred via TSE to the Department of Genetics at Reims University Hospital, designated to perform optical genome mapping while awaiting installation of the Saphyr scanner at Clermont-Ferrand University Hospital (DAN 2025 application).

Extraction, labeling, and imaging of long DNA molecules will be performed using the manufacturer's kits, following the provided instructions.

Results and Interpretation

Raw data will be analyzed and validated by cytogeneticists at Reims University Hospital using Bionano Access and Solve® software. Data will also be securely shared with the project lead, responsible for:

Performing a second independent analysis (with Bionano Access and Solve, available in the Cytogenetics Department), leveraging expertise acquired through participation in previous projects.

Providing final interpretation of results and disseminating clinically relevant findings for patient management.

Each sample will therefore benefit from dual review and dual expertise, ensuring the reliability of the results.

Parental segregation studies may be proposed to facilitate biological interpretation. If needed, collection of parental samples and consent procedures will be coordinated by the Department of Medical Genetics at Clermont-Ferrand University Hospital. Conclusive results will be communicated to the clinician who prescribed the WGS for patient management and genetic counselling.

ELIGIBILITY:
Inclusion Criteria

* Patients presenting with at least two congenital anomalies, with or without intellectual disability, and weighing more than 5 kg.
* Whole-genome sequencing performed by the AURAGEN laboratory deemed non-contributive (absence of class 4 or 5 variants, or identification of a VUS, or identification of only one variant in the context of a recessive disorder).
* Patient covered by a social security scheme.
* Patient able to understand and to oppose participation in the study.
* Written informed consent for genetic analyses, signed either by the patient or by their legal representatives (for minors), after clear and fair information about the study has been provided.

Non-Inclusion Criteria

* Patients for whom a non-genetic cause (infectious, environmental, or toxic) has been previously identified.
* Inability to obtain a compliant sample.
* Patient or holder of parental authority under guardianship or legal protection, deprived of liberty, or placed under court-ordered protection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
diagnostic yield of optical genome mapping (OGM) in multiple congenital anomalies with or without intellectual disability when whole-genome sequencing (WGS) is non-contributive | day 1 (inclusion and blood collection)
  Assessing the diagnostic yield of optical genome mapping (OGM) in multiple congenital anomalies with or without intellectual disability when whole-genome sequencing (WGS) is non-contributive (absence of causal genetic variation or detection of a variant of uncertain significance (VUS) or a single variant in a recessive disorder).

SECONDARY OUTCOMES:
Number of reclassified variants intially considered as VUS (Variants of Uncertain/Unknown Signification) | day 1 (inclusion and blood collection)
  Assessment of the number of variants initially classified as VUS (variants of uncertain/unknown significance) that were reclassified as benign or pathogenic variants
Number of patients in whom a new candidate gene/pathogenic mechanism is identified | day 1 (inclusion and blood collection)
Evaluation of the feasibility (duration) of the technique in current practice in 1st-line, 2nd-line (after routine tests such as chromosomal microarray, exome sequencing…), or 3rd-line in the case of non-contributive WGS based on several criteria | day 1 (inclusion and blood collection)
  Evaluation of technical duration (hours)
Evaluation of the feasibility of the technique (failure) in current practice in 1st-line, 2nd-line (after routine tests such as chromosomal microarray, exome sequencing…), or 3rd-line in the case of non-contributive WGS based on several criteria | day 1 (inclusion and blood collection)
  failure rate number
Evaluation of the feasibility of the technique (reprocessing) in current practice in 1st-line, 2nd-line (after routine tests such as chromosomal microarray, exome sequencing…), or 3rd-line in the case of non-contributive WGS based on several criteria | day 1 (inclusion and blood collection)
  reprocessing rate number
Evaluation of the feasibility of the technique (interpretation) in current practice in 1st-line, 2nd-line (after routine tests such as chromosomal microarray, exome sequencing…), or 3rd-line in the case of non-contributive WGS based on several criteria | day 1 (inclusion and blood collection)
  Evaluation of biological interpretation time (hours)
Assess the impact of using these new technologies on patient management. | day 1 (inclusion and blood collection)
  Percentage of patients for whom the OGM results led to a change in clinical management.

CONTACTS AND LOCATIONS:
Overall Officials: Lise LACLAUTRE, Study Chair — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No